CLINICAL TRIAL: NCT00122746
Title: Doctoral CRP on Clinical and Experimental Studies to Improve Radiotherapy Outcome in AIDS Cancer Patients
Brief Title: Clinical and Experimental Studies to Improve Radiotherapy Outcome in AIDS Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E33022
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Cancer of the Cervix
Keywords: Cervical Cancer; AIDS; External Beam Radiotherapy; Brachytherapy; Cisplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy alone (Active Comparator): EBRT pelvis 46 Gy, 4 field box technique + ICBT LDR 1x30 Gy/A or HDR 3x8 Gy/A
  Interventions: Radiation: Radiotherapy alone
- Radiotherapy plus Chemotherapy (Experimental): EBRT pelvis 46 Gy, 4 field box technique + ICBT LDR 1x30 Gy/A or HDR 3x8 Gy/A + weekly cisplatin 30 mg/m2 during EBRT
  Interventions: Radiation: Radiotherapy with cisplatin

INTERVENTIONS:
Radiation: Radiotherapy alone — EBRT pelvis 46 Gy 4 field box technique + ICBT LDR 1x30 Gy/A or HDR 3x8 Gy/A
  Arms: Radiotherapy alone
Radiation: Radiotherapy with cisplatin — EBRT pelvis 46 Gy 4 field box technique + ICBT LDR 1x30 Gy/A or HDR 3x8 Gy/A + weekly cisplatin 30 mg/m2 during EBRT
  Arms: Radiotherapy plus Chemotherapy

SUMMARY:
The researchers plan:

* To undertake clinical studies of radiotherapy with or without the administration of the chemotherapeutic agent cisplatin, known to be a radiosensitizer;
* To perform pre-clinical studies of the radiosensitivity of human fibroblasts and cervical cancer cell lines in culture, with or without the addition of various HIV proteins or protease inhibitors, in order to determine the extent of any cellular radiosensitizing properties of these molecules;
* To develop strategies for sensitizing tumour cells to radiation, specifically by down-regulating specific viral proteins that are known to be factors associated with resistance to radiotherapy.

DETAILED DESCRIPTION:
Clinical study addresses the question of whether radiotherapy plus weekly cisplatin offers an advantage over the same radiotherapy given alone in AIDS patients with cervix cancer. External beam radiotherapy is used with 50 Gy in 25 daily fractions (last interim analysis, October 2005) suggested lowering the total dose down to 46 Gy in 23 daily fractions). Brachytherapy component was specified as either 30 Gy of LDR in a single fraction or 3 fractions of 8 Gy using HDR. Cisplatin was administered weekly at a dose of 30 mg/sqm.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the cervix
* AIDS

Exclusion Criteria:

* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Estimated)
Dates: Start 2004-12; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
3 year recurrence free survival | 3 years

SECONDARY OUTCOMES:
Incidence of Grade 3 acute toxicity | 3 months
Pelvic control rates | 3 years
Tumour response at 3 months. | 3 months
Cancer specific survival rates. | 3 years
Overall survival rates. | 3 years
Acute and late toxicities after the treatment. | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo H. Zubizarreta, M.D., Study Director — International Atomic Energy Agency
Locations (5):
- Dept. of Atomic Energy, Tata Memorial Centre, Mumbai, India
- Johannesburg Hospital, Johannesburg, South Africa
- Ocean Road Cancer Institute, Dar es Salaam, Tanzania
- Radiotherapy Centre, Kampala, Uganda
- Radiotherapy Centre, Harare, Zimbabwe

REFERENCES:
- See also: International Atomic Energy Agency. Research Contracts Administration — http://www.iaea.org